## Data Analysis Plan for a pilot feasibility study of providing substance use treatment in the Black Church

PI: Ayana Jordan MD, PhD Data Manager: Theresa Babuscio

Updated 12/3/2020

This study is being conducted to determine the feasibility of recruiting Black adults with substance use disorder from within the Black Church and immediate surrounding community and retaining them in treatment, within a church setting.

A consort diagram will be used to assess the flow of participants from screening through week 8. Since this is a single arm trial cross tabs and ANOVA's will be run to describe the sample on characteristics such as age, sex, education, marital status.

 We will measure acceptability of treatment by giving each participant a post-intervention satisfaction survey as well as a qualitative exit interview, to fully assesses satisfaction with the intervention, perception of outcome, attitudes about spiritual practices accompanying CBT modules, and whether the participant would recommend this program to a friend.

This will be done by calculating the mean and standard deviation of each question.

2. Feasibility will be measured by at least 2/3 of participants (N=27) completing the CBT4CBT intervention.

This will be a done by calculating the mean and standard deviation of number of sessions attended over the 8-week trial.

3. Secondary analyses will include significant reductions in drug use, as measured by mean change scores in the severity and quantity of substance use, and functioning over the course of treatment intervention.

As the study was implemented this outcome was refined to better reflect the aims of the study (recruiting and retention participants in treatment). A change score will not be calculated.